CLINICAL TRIAL: NCT01173445
Title: A Pilot Study on the Assessment of Circulating Tumors Cells and Circulating Endothelial Cells in Renal Cell Carcinoma
Brief Title: Circulating Tumors Cells and Circulating Endothelial Cells in Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 12203
Record Dates: First submitted 2010-07-27; First posted 2010-08-02 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Renal Cell Carcinoma
Keywords: cancer; kidney; renal cell; tumor cells; circulating tumor cells; circulating endothelial cells
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples will be collected at the following times:
  * one draw prior to treatment initiation
  * one draw after completion of two treatment cycles
  * one draw at the time of disease progression
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to see if researchers can detect circulating tumor cells (CTC) and circulating endothelial cells (CEC) in the blood.

DETAILED DESCRIPTION:
Circulating tumors cells (CTCs) and circulating endothelial cells (CECs) are found in the peripheral blood of most common malignancies and are promising surrogate biomarkers. The CellSearchTM CTC assay is currently approved by the Food and Drug Administration as an adjunct for monitoring disease status in breast, prostate and colon carcinomas; and evidence in breast cancer suggests that CTCs are an independent predictor of overall survival and progression-free survival. Evolving data demonstrates a potential role of CTCs as a surrogate assessment for treatment response. The benefit of this approach in renal cell cancer(RCC) is unknown and further investigation is needed to determine the feasibility of using the CellSearchTM CTC Assay in this malignancy.

Circulating endothelial cells (CECs) are increased in the peripheral blood of cancer patients and appear to be a marker of tumor related angiogenesis. Studies suggest that CECs increase in the setting of progressive disease and decrease in response to treatment with an antiangiogenic agent. Although current data evaluating CECs in RCC is limited, there is significant interest in CEC evaluation as a marker of treatment response given the majority of current FDA approved RCC therapies target tumor angiogenesis.

The overall objective of this protocol is to obtain preliminary data and experience using our Cell Search Assay system which can be used for future grant applications. Our hypothesis is that CTCs and/or CECs will be valuable and versatile biomarkers for therapeutic response, determination of relapse and survival in patients with renal cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with radiographic or histologic evidence of renal cell carcinoma who is scheduled to begin treatment with one of the following antiangiogenic agents: sunitinib, sorafenib, temsirolimus or bevacizumab.
* Patients must be candidates to be treated with one of the above agents but there is no limit on the number of prior therapies (i.e. first line or subsequent treatment setting).
* Patients scheduled to undergo debulking nephrectomy prior to beginning systemic therapy do not require histologic diagnosis prior to baseline testing.
* Must be able and willing to sign informed consent.
* Patients must be 18 years or older.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be approached for participation during regular Cancer Center clinic visits.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Determine if the number of CTCs and CECs in subject's blood changes with treatment. | Pre-nephrectomy subjects - one week prior to beginning treatment and at first planned radiologic assessment. Other subjects will be collected at baseline and at time of first radiograph assessment of response.
  Subject samples will be used to see if CTCs and/or CECs will be valuable and versatile biomarkers for therapeutic response, determination of relapse and survival in patients with renal cell cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J VanVeldhuizen, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States